CLINICAL TRIAL: NCT02226211
Title: Ambu® Aura-iTM Laryngeal Mask Versus Air-QTM Intubating Laryngeal Airway as Conduits for Tracheal Intubation in Adults. A Randomized Comparative Clinical Trial
Brief Title: Ambu Aura-i Laryngeal Mask Versus Air-Q Intubating Laryngeal Airway for Tracheal Intubation in Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: N-46-2014
Record Dates: First submitted 2014-08-22; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Failed or Difficult Intubation (Anaesthesia Complications)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- air-Q group (Experimental)
  Interventions: Device: Air-Q intubation laryngeal airway
- aura-i group (Experimental)
  Interventions: Device: Ambu-Aura i laryngeal mask

INTERVENTIONS:
Device: Air-Q intubation laryngeal airway — The size selection of the air-Q ILA will follow the manufacture guideline to be size 3.5 for females and size 4.5 for males After induction of general anesthesia, the devices will be inserted by using midline insertion technique, then cuff will be inflated according to manufacture recommendations.
  After successful insertion of the air-Q, the appropriate endoracheal tube (ETT) will be loaded over the fiberoptic bronchoscopy, and the connector will be removed too. The bronchoscope will be introduced and advanced throughout the airway tube to just proximal to ventilating orifice, a video image of the fiberoptic view will be recorded and saved on CD to be graded later by an independent observe. The fiberoptic then will be advanced and once the carina is seen, the ETT is will be slided into the trachea.
  After successful intubation, the device will be removed according to the manufactures guides using removal stylet .
  Arms: air-Q group
Device: Ambu-Aura i laryngeal mask — The size selection of the device will follow the manufacture guideline according to the patient weight, size 4 for (50-70kg), size 5 (70-100) and size 6 (> 100kg).
  After induction of general anesthesia, the devices will be inserted by using midline insertion technique, then cuff will be inflated according to manufacture recommendations.
  After successful insertion of the aura-i, the appropriate endoracheal tube (ETT) will be loaded over the fiberoptic bronchoscopy, and the connector will be removed too. The bronchoscope will be introduced and advanced throughout the airway tube to just proximal to ventilating orifice, a video image of the fiberoptic view will be recorded and saved on CD to be graded later by an independent observe. The fiberoptic then will be advanced and once the carina is seen, the ETT is will be slided into the trachea.
  After successful intubation, the device will be removed according to the manufactures guides using another ETT.
  Arms: aura-i group

SUMMARY:
Supraglottic airway devices (SGA) become a routine part of the daily anesthesia practice. they can be used as primary airway devices or as conduits for endoracheal intubation and they become an integral part in the recent guidelines for managing difficult airway.

Air-Q ILA has been used successfully as 1ry airway and also as a conduits for endotracheal intubation.

The Ambu® Aura-i TM laryngeal mask is a new disposable SGA claimed to have special advantage over the competitors but not will studied as a conduit for endoracheal intubation.

This study is designed to compare the performance of Ambu®Aura-i™ laryngeal mask with the air-Q ILA as conduits for fiberoptic-guided tracheal intubation in adult population.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18-60 years old, ASA I and II and scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* history of cardiopulmonary disease, gastro-esophageal reflux disease, abnormal airway anatomy, body mass index > 30 kg.m-2, surgical procedures including head and neck or performed in position other than supine or lithotomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
duration of fiberoptic guided insertion of the ETT through the device | duration of induction of general anesthesia, an expected average of 20 minutes. and it is the time span between disconnection of the breathing circuit from the device till reconnection to the ETT and appearance of 1st capnogram wave.

SECONDARY OUTCOMES:
duration of device insertion | duration of induction of general anesthesia, an expected average of 20 minutes and it is the time span between removal of the face mask till device insertion and the chest rise seen after two consecutive positive pressure manual breaths.
Time of device removal | duration of induction of general anesthesia, an expected average of 20 minutes, and it is the time span between disconnection of the breathing circuit from ETT and reconnection to ETT after device removal with appearance of the 1st capnogram wave.
number of insertion attempts | duration of induction of general anesthesia, an expected average of 20 minutes and it is the time span from removal of face mask till complete insertion or failed third insertion trial of the device
complication during the procedure | average of 20 minutes after induction of general anesthesia, it is the time from removal of face mask, till removal of the device and appearance of the first wave on the capnogram
vital sign in form of mean arterial blood pressure, heart rate and oxygen saturation | average of 20 minutes, and it is the time from time of induction of general anesthesia til completion of endotracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of Medicine - Cairo university, Cairo, Cairo Governorate, Egypt